CLINICAL TRIAL: NCT02272244
Title: Increasing Colorectal Cancer (CRC) Screening Among Hispanic Primary Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Lehigh Valley Hospital (Other); Fox Chase Cancer Center (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AD-1306-01882; JT 5992 (Other: JeffTrial Number)
Record Dates: First submitted 2014-10-20; First posted 2014-10-22 (Estimated); Results first posted 2019-08-12 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; Cancer Screening; Decision Support; Navigation
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard (Active Comparator): SI Group participants will be mailed a set of standard materials. The materials will include a letter from the participant's primary care practice encouraging selection and performance of either (1) colonoscopy screening, or (2) stool blood test (SBT) screening. Accompanying the letter will be instructions for arranging a colonoscopy appointment and instructions for completing an enclosed immunochemical SBT kit. Print materials and contacts will be provided, in both English and Spanish, after the baseline survey. At 45 days following random assignment that encourages screening.
  Interventions: Behavioral: Standard
- Decision Support & Navigation (Experimental): DSNI Group will be mailed print materials, including a letter from the practice on CRC screening, an informational booklet, and instructions for arranging a colonoscopy appointment and for completing an enclosed immunochemical SBT kit. All materials will be provided in both English and Spanish. Within 7 days after this mailing, participants will receive a telephone call from a trained bilingual study navigator. Following the call, the navigator will enter the participant's screening plan into the participant's electronic medical record, send the participant a letter describing the screening plan, and send the participant's primary care provider a copy of that same letter. At 45 days following random assignment, research staff will send participants a reminder letter encouraging the participant's preferred test. At 6 months after randomization, the navigator will send the provider and their office manager a participant CRC screening status report.
  Interventions: Behavioral: Decision Support & Navigation

INTERVENTIONS:
Behavioral: Decision Support & Navigation
  Arms: Decision Support & Navigation
Behavioral: Standard
  Arms: Standard

SUMMARY:
This study is designed to test a standard mailed intervention (SI) versus a novel decision support and navigation intervention (DSNI). Working with patients and stakeholders, this randomized trial will include 400 Hispanic men and women who are 50 to 75 years of age, patients in community based primary care practices, and are eligible for CRC screening. We will consent, survey, and randomize participants either to the SI Group (n=200) or the DSNI Group (n=200). Study specific aims are to: (1) Assess intervention (DSNI versus SI) impact on overall CRC screening adherence; (2)Assess intervention (DNSI versus SI) impact on CRC screening decision stage; (3) Assess intervention (DNSI versus SI) impact on test-specific CRC screening adherence; and (4) Assess intervention (DNSI versus SI) impact on CRC and knowledge and perceptions.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Self-identifies as being Hispanic or Latino
* 50 to 75 years of age

Exclusion Criteria:

* Previous diagnosis of CRC
* Up to date with CRC screening guidelines.
* Personal history of inflammatory bowel disease
* Personal history of polyps
* Family history of CRC diagnosed before the age of 60 years

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2014-10-01; Primary Completion 2017-01-20 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald E Myers, PhD, Principal Investigator — Thomas Jefferson University
Locations (3):
- United States (3):
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Myers RE, Stello B, Daskalakis C, Sifri R, Gonzalez ET, DiCarlo M, Johnson MB, Hegarty SE, Shaak K, Rivera A, Gordils-Molina L, Petrich A, Careyva B, de-Ortiz R, Diaz L. Decision Support and Navigation to Increase Colorectal Cancer Screening Among Hispanic Patients. Cancer Epidemiol Biomarkers Prev. 2019 Feb;28(2):384-391. doi: 10.1158/1055-9965.EPI-18-0260. Epub 2018 Oct 17. PMID 30333221

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2,720 study invitation letters sent to subjects from 5 practices that appeared to meet eligibility criteria based on medical records.
Pre-assignment Details: 2,320 were excluded
  * 98 contact not attempted (recruitment goals met or known ineligible)
  * 504 were determined up to date on screening
  * 182 were ineligible for other reasons
  * 256 refused
  * 717 were unable to be contacted
  * 563 were wrong numbers
Period: Overall Study
Arm/Group | Standard | Decision Support & Navigation
Started | 203 | 197
Completed | 203 | 197
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard: SI Group participants will be mailed a set of standard materials. The materials will include a letter from the participant's primary care practice encouraging selection and performance of either (1) colonoscopy screening, or (2) stool blood test (SBT) screening. Accompanying the letter will be instructions for arranging a colonoscopy appointment and instructions for completing an enclosed immunochemical SBT kit. Print materials and contacts will be provided, in both English and Spanish, after the baseline survey. At 45 days following random assignment that encourages screening.
  Standard
- Decision Support & Navigation: DSNI Group will be mailed print materials, including a letter from the practice on CRC screening, an informational booklet, and instructions for arranging a colonoscopy appointment and for completing an enclosed immunochemical SBT kit. All materials will be provided in both English and Spanish. Within 7 days after this mailing, participants will receive a telephone call from a trained bilingual study navigator. Following the call, the navigator will enter the participant's screening plan into the participant's electronic medical record, send the participant a letter describing the screening plan, and send the participant's primary care provider a copy of that same letter. At 45 days following random assignment, research staff will send participants a reminder letter encouraging the participant's preferred test. At 6 months after randomization, the navigator will send the provider and their office manager a participant CRC screening status report.
  Decision Support & Navigation
- Total: Total of all reporting groups
Arm/Group | Standard | Decision Support & Navigation | Total
Number analyzed (Participants) | 203 | 197 | 400
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (6.5) | 57.2 (6.4) | 57.3 (6.5)
Age, Customized [Count of Participants; unit: Participants]
  Age (years): 50-59 | 140 | 137 | 277
  Age (years): 60-69 | 47 | 48 | 95
  Age (years): 70-79 | 16 | 12 | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 117 | 235
  Male | 85 | 80 | 165
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White/Caucasian | 64 | 69 | 133
  Race: Black/African American | 61 | 57 | 118
  Race: Other | 42 | 49 | 91
  Race: Unknown/Not Reported | 36 | 22 | 58
Marital Status [Count of Participants; unit: Participants]
  Married | 94 | 78 | 172
  Living as marreid | 10 | 10 | 20
  Divorced | 25 | 26 | 51
  Separated | 20 | 13 | 33
  Widowed | 7 | 17 | 24
  Never married | 47 | 53 | 100
Education [Count of Participants; unit: Participants]
  Less than HS | 90 | 102 | 192
  HS/GED | 58 | 51 | 109
  Completed Non-College/Business/Trade/Tech | 13 | 8 | 21
  2-yr Associates | 16 | 19 | 35
  College Degree and above | 26 | 17 | 43
Employment Status [Count of Participants; unit: Participants]
  Working full-time | 44 | 41 | 85
  Working part-time | 41 | 35 | 76
  Keeping House | 45 | 45 | 90
  Unable to Work/Disability | 53 | 62 | 115
  Retired | 20 | 14 | 34
Family Income [Count of Participants; unit: Participants]
  Under $14,999 | 144 | 136 | 280
  $15,000-$29,000 | 37 | 45 | 82
  $30,000-$45,999 | 18 | 12 | 30
  $46,000-$59,999 | 3 | 4 | 7
  Unknown/Not Reported | 1 | 0 | 1
Insurance Status [Count of Participants; unit: Participants]
  Insured | 140 | 141 | 281
  Uninsured | 58 | 53 | 111
  Unknown/Not Reported | 5 | 3 | 8
Help Reading Materials from Doctor [Count of Participants; unit: Participants]
  Never | 94 | 96 | 190
  Rarely | 16 | 15 | 31
  Sometimes | 45 | 44 | 89
  Often | 11 | 10 | 21
  Always | 37 | 32 | 69
Practice [Count of Participants; unit: Participants]
  Centro de Salud | 40 | 43 | 83
  Lehigh Valley Family Health Center | 47 | 45 | 92
  Lehigh Valley Physician's Practice | 76 | 74 | 150
  AIDS Activity Office | 10 | 10 | 20
  Neighborhood Health Center of the Lehigh Valley | 30 | 25 | 55
Years in the US [Count of Participants; unit: Participants]
  Less than 1 year | 1 | 0 | 1
  1-3 | 9 | 12 | 21
  4-6 | 12 | 13 | 25
  7-10 | 11 | 18 | 29
  More than 10 | 145 | 132 | 277
  Born in the US | 24 | 22 | 46
  Unknown | 1 | 0 | 1
Region of Birth [Count of Participants; unit: Participants]
  United States | 24 | 22 | 46
  Caribbean- Puerto Rico | 81 | 79 | 160
  Caribbean- Dominican Republic and Cuba | 65 | 63 | 128
  Central America/Mexico | 19 | 18 | 37
  South America | 14 | 15 | 29
Language Most Spoken at Home [Count of Participants; unit: Participants]
  Spanish | 163 | 168 | 331
  Both | 26 | 15 | 41
  English | 14 | 14 | 28
Language Score [Mean (Standard Deviation); unit: units on a scale] — 4-item Likert-type scale with scores that can range from 1-5 with 1 indicating more English used and 5 indicating Spanish used
  units on a scale | 4.28 (1.05) | 4.38 (1.00) | 4.33 (1.02)
Preferred CRC screening test [Count of Participants; unit: Participants]
  Stool Blood Test | 53 | 33 | 86
  Even | 133 | 142 | 275
  Colonoscopy | 17 | 22 | 39
CRC screening decision stage [Count of Participants; unit: Participants]
  Decided not to do | 2 | 2 | 4
  Not considering | 7 | 2 | 9
  Haven't decided | 20 | 27 | 47
  Decided to do | 174 | 166 | 340

OUTCOME MEASURES:

1. Primary Outcome: Overall Screening Adherence
Description: The two study groups will be compared in terms of the fraction of participants who undergo CRC screening (through SBT, colonoscopy, flexible sigmoidoscopy, etc.) within 12 months of the randomization date. Screening will be measured using data from the 6-month survey and the 12-month chart audit.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard | Decision Support & Navigation
Number analyzed (Participants) | 203 | 197
Participants
  Screened | 88 | 153
  Not Screened | 115 | 44
Statistical Analysis 1: Comparison: Standard vs Decision Support & Navigation; Test type: Superiority; p < 0.001, Regression, Logistic; Model adjusted for age, sex, practice, baseline preferred test and baseline overall decision stage; Odds Ratio (OR) = 4.83, 95% CI 2-sided [3.08 to 7.58]

2. Secondary Outcome: Change in Screening Decision Stage
Description: At baseline and endpoint (6-month) survey, participants were asked about their decision stage regarding CRC screening. Possible decision stages are, ranked from lowest to highest stage: Decided not to do, Not considering, Haven't decided, Decided to Do and Done, with "Done" only possible at endpoint.
Time Frame: 6 months
Population: Participants with complete baseline and endpoint survey data
Measure: Count of Participants; unit: Participants
Arm/Group | Standard | Decision Support & Navigation
Number analyzed (Participants) | 123 | 123
Participants
  Forward Change | 61 | 97
  No Change | 52 | 23
  Backward Change | 10 | 3
Statistical Analysis 1: Comparison: Standard vs Decision Support & Navigation; Test type: Superiority; p < 0.001, Regression, Logistic; Model compares Forward Change to No Change or Backwards Change and is adjusted for all baseline covariates; Odds Ratio (OR) = 4.91, 95% CI 2-sided [2.55 to 9.47]

3. Secondary Outcome: Test Specific Screening Adherence
Description: Test adherence (SBT or endoscopy) will be assessed using 6-month survey and 12-month medical records data. The two study groups will be compared in terms of the fraction of participants who have a screening test within 12 months.
Time Frame: 12 Months
Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard | Decision Support & Navigation
Number analyzed (Participants) | 203 | 197
Participants
  None | 115 | 44
  Stool Blood Test | 76 | 113
  Colonoscopy | 12 | 40
Statistical Analysis 1: Comparison: Standard vs Decision Support & Navigation; Test type: Superiority; p < 0.001, Regression, Multinomial; Model compared rates of SBT, CX and none; model is adjusted for age, sex, practice, baseline preferred test and baseline overall decision stage; Reference for the outcome is No Screening; reference for the study group is the Standard Intervention group
Statistical Analysis 2: Comparison: Standard vs Decision Support & Navigation; Test type: Superiority; p = 0.001, Odds Ratio (OR); Stool Blood Test vs None; Odds Ratio (OR) = 4.20, 95% CI 2-sided [2.63 to 6.70]
Statistical Analysis 3: Comparison: Standard vs Decision Support & Navigation; Test type: Superiority — Colonscopy vs None; p = 0.001, Odds Ratio (OR); Odds Ratio (OR) = 8.79, 95% CI 2-sided [4.13 to 18.74]

4. Secondary Outcome: Screening Knowledge and Perceptions
Description: Knowledge and perceptions (Preventive Health Model scales) about CRC and screening will be assessed in a 6-month survey. Knowledge was measured by a set of 10 true-false statements about CRC and CRC screening. Knowledge was scored as the number of items correct with a possible range of 0 to 10. Perceptions about CRC and screening were measured using a 20-item scale based on the Preventive Health Model. Items were measured on a 5 point Likert scale ranging from 1 = Strongly Disagree to 5 = Strongly Agree. The total score and subscale scores were computed by taking the mean of component items resulting in scores that could range from 1 to 5, with higher scores indicating more favorable attitudes towards the CRC screening preventive health behavior.
Time Frame: 6 months
Population: Participants with complete baseline and 6-month survey data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard | Decision Support & Navigation
Number analyzed (Participants) | 122 | 123
units on a scale
  Preventive Health Model (PHM) | 3.8 (0.5) | 3.8 (0.6)
  PHM: Salience | 4.8 (0.5) | 4.7 (0.6)
  PHM: Response Efficacy | 4.5 (0.7) | 4.5 (0.7)
  PHM: Susceptibility | 2.6 (1.0) | 2.8 (1.0)
  PHM: Worries and Concerns | 3.1 (1.1) | 3.1 (1.1)
  PHM: Social Support and Influence | 4.4 (0.8) | 4.4 (0.9)
  Knowledge Test | 4.7 (1.8) | 4.6 (2.1)
Statistical Analysis 1: Comparison: Standard vs Decision Support & Navigation; Test type: Superiority; p = 0.862, Regression, Linear; Model of difference in Preventive Health Model (PHM) total score adjusts for all baseline covariates; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.15 to 0.13] — Model compares DSNI to SI
Statistical Analysis 2: Comparison: Standard vs Decision Support & Navigation; Test type: Superiority; p = 0.880, Regression, Linear; Model of knowledge test score adjusts for all baseline covariates; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-.47 to .55] — Model compares DSNI to SI

ADVERSE EVENTS:
Time Frame: 1 Year from baseline
Arm/Group | Standard | Decision Support & Navigation
All-Cause Mortality (participants affected / at risk) | 0/203 | 0/197
Serious Adverse Events (participants affected / at risk) | 0/203 | 0/197
Other Adverse Events (participants affected / at risk) | 0/203 | 0/197

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-14): https://cdn.clinicaltrials.gov/large-docs/44/NCT02272244/Prot_SAP_000.pdf